CLINICAL TRIAL: NCT02134210
Title: A Double-Blind, Randomized, Parallel-Group, Active-Control Study to Compare the Efficacy and Safety of CHS-0214 Versus Enbrel in Subjects With Chronic Plaque Psoriasis (RaPsOdy)
Brief Title: Comparison of CHS-0214 to Enbrel (Etanercept) in Patients With Chronic Plaque Psoriasis (PsO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS-0214-04
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Plaque Psoriasis
Keywords: PsO
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enbrel (etanercept) (Active Comparator): Enbrel 50mg twice weekly times 12 weeks
  Interventions: Drug: Etanercept
- CHS-0214 (Experimental): CHS-0214 50mg twice weekly times 12 weeks
  Interventions: Drug: CHS-0214

INTERVENTIONS:
Drug: Etanercept — Head-to-head comparison
  Other Names: Enbrel; European Enbrel
  Arms: Enbrel (etanercept)
Drug: CHS-0214
  Arms: CHS-0214

SUMMARY:
This is a two part study comparing CHS-0214 to Enbrel in patients with chronic plaque PsO who have not yet received any biologic therapy for any indication (other than insulin or hormones).

DETAILED DESCRIPTION:
Pt. 1 is a 12-week randomized, double-blind, active-control, parallel-group, multi-center global study. The primary end point is 75% improvement from baseline according to the Psoriasis Area and Severity Index (PASI-75). Comparing CHS-0214 to Enbrel for efficacy and safety at a dosage of 50mg subcutaneous (Sc) twice weekly.

Pt. 2 is a 40-week randomized, double-blind, active-control, parallel-group, multi-center global study where CHS-0214 and Enbrel dosage is reduced to 50mg Sc weekly for maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* PsO diagnosis for 6 months
* Active disease: PASI greater than or equal to 12, Physician's Static Global Assessment (PSGA) score greater than or equal to 3 (based on a scale or 0-5),
* Body Surface Area (BSA) involved with PsO greater than or equal to 10%
* Dermatology Life Quality Index (DQLI) greater than or equal to 10
* Previously received phototherapy or systemic non-biologic therapy for PsO

Exclusion Criteria:

* Forms of Psoriasis other than PsO
* Drug induced Psoriasis
* Positive QuantiFERON-tuberculosis (TB) Gold Test
* Presence of significant comorbid conditions
* Chemistry and hematology values outside protocol specified range
* Major systemic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Finck, M.D., Study Director — Coherus Oncology, Inc.
Locations (100):
- United States (50):
  - Arizona Research Center, Phoenix, Arizona
  - Radiant Research - Scottsdale, Scottsdale, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Dream Team Clinical Research, Anaheim, California
  - Private Practice, Encino, California
  - Kaiser Permanente, Los Angeles, California
  - Skin Surgery Medical Group, Inc, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Healthcare Partners Medical Group, Torrance, California
  - Horizons Clinical Research Center, Denver, Colorado
  - The Savin Center, New Haven, Connecticut
  - New England Research Associates, Trumbull, Connecticut
  - Florida Academic Dermatology Center (U of Miami Hospital), Miami, Florida
  - Radiant Research - Pinellas Park, Pinellas Park, Florida
  - Atlantic Clinical Research Collaborative, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Radiant Research - Atlanta, Atlanta, Georgia
  - Private Practice - Jamie Weisman, Atlanta, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Springfield Clinic, Springfield, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, Overland Park, Kansas
  - Derm Research, Louisville, Kentucky
  - Hamzavi Dermatology Clinical Research, Fort Gratiot, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Radiant Research - Edina, Edina, Minnesota
  - Central Dermatology, St Louis, Missouri
  - The Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Skin Search of Rochester, Inc, Rochester, New York
  - DermResearch Center of New York, Stony Brook, New York
  - PMG Research of Carey, LLC, Cary, North Carolina
  - DJL Clinical Research, Charlotte, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clincal Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Radiant Research - Anderson, Anderson, South Carolina
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - Radient Research - Greer, Greer, South Carolina
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Neighborhood Medical Center, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Heights Dermatology and Aesthetic Center, Houston, Texas
  - Progressive Clinical Research - San Antonio, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Associates, PLLC, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Australia (5):
  - Woden Dermatology Pty, Phillip, Australian Capital Territory
  - Dr S P Shumack (St George Dermatology and Skin Cancer Center), Kogarah, New South Wales
  - Dr S P Shumack (Central Sydney Dermatology), Sydney, New South Wales
  - North Eastern Health Specialists, Hectorville, South Australia
  - Sinclair Dermatology, East Melbourne, Victoria
- Canada (10):
  - E and D Woolner Professional Corporation, Calgary, Alberta
  - Institute for Skin Advancement Inc, Calgary, Alberta
  - CCA Medical Research Corporation, Ajax, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - North Bay Dermatology Centre Inc, North Bay, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - SKiN Center for Dermatology, Peterborough, Ontario
  - Private Practice, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research Inc, Waterloo, Ontario
- Germany (6):
  - MVZ Reichenberger Str., Aerztehaus "Rudolf Virchow, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Hautklinik Universitaetsklinikum Erlangen, Erlangen
  - Johann Wolfgang Hospital - Goethe University, Frankfurt
  - Dermatologikum Hamburg, Hamburg
  - University Hospital Schleswig-Holstein - Campus Luebeck, Lübeck
- Israel (4):
  - Haemek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Poland (18):
  - NZOZ Osteo-Medic s.c. Artur Racewicz, Jerzy Supronik, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Osteoporozy i Chorób Kostno-Stawowych J. Badurski S.J, Bialystok
  - Centrum Badan Klinicznych PI-House Sp. Z o.o, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Specjalistyczny Osrodek ALL-MED, Krakow
  - Krakowskie Centrum Medyczne, Krakow
  - Center Med, Krakow
  - Specjalistyczne Gabinety Lekarskie "Dermed, Lodz
  - Centrum Medyczne SYNEXUS POZNAN, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - SANUS Szpital Specjalistyczny Sp. z o.o, Stalowa Wola
  - EuroMedis Sp. z o.o., Szczecin
  - NZOZ "Nasz Lekarz" Praktyka Grupowa Lekarzy z Przychodnia Specjalistyczna, Torun
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Synexus Polska sp. z o.o, Wroclaw
  - Dermmedica Sp. z o.o, Wroclaw
- South Africa (7):
  - Vincent Pallotti Hospital, Pinelands, Cape Town
  - Synopsis Research, Rondebosch, Cape Town
  - Jongaie Research, Pretoria West, Pretoria
  - Helderberg Clinical Trial Centre, Somerset West, Western Cape
  - Dr IC Louw, Cape Town
  - Winelands Rheumatology Centre, Stellenbosch
  - Clinical Projects Research, Worcester

RESULTS

PARTICIPANT FLOW:
Groups:
- CHS-0214: CHS-0214 50mg twice weekly times 12 weeks
  CHS-0214
Period: Part One: Weeks 0-12
Arm/Group | Enbrel (Etanercept) | CHS-0214
Started | 260 | 261
Completed | 241 | 255
Not Completed | 19 | 6
Period: Part Two: Weeks 13-48
Arm/Group | Enbrel (Etanercept) | CHS-0214
Started | 241 | 255
Completed | 211 | 227
Not Completed | 30 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enbrel (Etanercept) | CHS-0214 | Total
Number analyzed (Participants) | 260 | 261 | 521
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.75) | 44.3 (12.86) | 43.7 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 156
  Male | 180 | 185 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 240 | 241 | 481
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 4 | 6
  White | 236 | 242 | 478
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving PASI-75(75% Improvement in Psoriasis Area and Severity Index) From Baseline at Week 12
Description: The Psoriasis Area and Severity Index (PASI) is well established in the medical literature and is internationally the most widely used instrument to assess the severity of Psoriasis.
  Proportion of subjects achieving PASI-75 from baseline at Week 12. This was the primary endpoint supporting a Biologics Licensing Application in the US.
Time Frame: 12-weeks
Measure: Number; unit: participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
participants | 142 | 147

2. Primary Outcome: Mean Percent Change in PASI (Psoriasis Area and Severity Index) at 12 Weeks
Description: Mean percent changed in PASI from baseline (last non-missing value prior to first dose) at Week 12. This was the primary endpoint supporting the Marketing Authorization Application in the EU.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 226 | 228
percentage of change | -73.4 (25.0) | -76.7 (21.1)

3. Secondary Outcome: Mean Percent Change in PASI (Psoriasis Area and Severity Index) From Baseline
Description: Mean percent change in PASI from baseline at Weeks 4, 8, 12, 24, 36, and 48
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Population: Part 2 of the study took place from week 13-48 and not all subjects that started the study were included in analysis
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
percentage of change
  Week 4 | -42.1 (24.93) | -43.2 (22.63)
  Week 8 | -62.8 (24.23) | -65.7 (22.16)
  Week 12 | -76.0 (21.96) | -77.0 (20.74)
  Week 24: number analyzed (Participants) | 213 | 225
  Week 24 | -83.3 (17.5) | -80.8 (20.43)
  Week 36: number analyzed (Participants) | 213 | 225
  Week 36 | -82.8 (20.44) | -81.9 (18.55)
  Week 48: number analyzed (Participants) | 213 | 225
  Week 48 | 82.9 (18.55) | -80.9 (25.08)

4. Secondary Outcome: Number of Participants Who Achieved PASI - 75 (75% Improvement in Psoriasis Area and Severity Index)
Description: The proportion of subjects who achieved PASI-75 (75% Improvement in Psoriasis Area and Severity Index) from baseline at Weeks 4, 8, 12, 24, 36, and 48.
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Measure: Count of Participants; unit: Participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 260 | 261
Participants
  Week 4 | 221 | 228
  Week 8 | 213 | 225
  Week 12 | 213 | 225
  Week 24 | 204 | 221
  Week 36 | 195 | 211
  Week 48 | 178 | 203

5. Secondary Outcome: Number of Subjects Who Achieved a 50% Improvement in Psoriasis Area and Severity Index (PASI-50) and a 90% Improvement in PASI (PASI-90)
Description: The proportion of subjects who achieved a 50% improvement in Psoriasis Area and Severity Index (PASI-50) and a 90% improvement in PASI (PASI-90) response rates from baseline at Weeks 4, 8, 12, 24, 36, and 48
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Measure: Number; unit: participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
participants
  Week 4 PASI-50 | 86 | 89
  Week 4 PASI-90 | 8 | 6
  Week 8 PASI-50 | 155 | 173
  Week 8 PASI-90 | 25 | 28
  Week 12 PASI-50 | 184 | 200
  Week 12 PASI-90 | 57 | 69
  Week 24 PASI-50 | 194 | 201
  Week 24 PASI-90 | 89 | 99
  Week 36 PASI-50 | 183 | 197
  Week 36 PASI-90 | 92 | 93
  Week 48 PASI-50 | 169 | 189
  Week 48 PASI-90 | 81 | 91

6. Secondary Outcome: Change in PSGA (Physician's Static Global Assessment) of Disease Activity on a Scale of 0 to 5
Description: Change in PSGA (Physician's Static Global Assessment) of disease activity on a scale of 0 to 5 from baseline to Weeks 4, 8, 12, 24, 36, and 48.
  Minimum Value: 0 Maximum Value: 5
  The PSGA of PsO (Psoriasis) was assessed on a scale of 0 to 5, with 0 indicating no PsO (clear of disease),1 (almost clear), and 2 or higher scores indicating more severe disease. Subjects with a clear (0) or almost clear (1) evaluation were considered PSGA responders.
Time Frame: 4, 8, 12, 24, 36, and 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
score on a scale
  Week 4 | -1.2 (0.83) | -1.2 (0.81)
  Week 8 | -1.8 (0.94) | -1.17 (0.88)
  Week 12 | -2.1 (1.05) | -2.1 (0.97)
  Week 24 | -2.2 (1.5) | -2.2 (1.07)
  Week 36 | -2.2 (1.17) | -2.1 (1.10)
  Week 48 | -2.1 (1.11) | -2.1 (1.15)

7. Secondary Outcome: The Proportion of Subjects With a Change in a PSGA (Physician's Static Global Assessment) Score = 0 to 1
Description: The proportion of subjects with a change in a PSGA (Physician's Static Global Assessment) score = 0 to 1, demonstrating clear or almost clear skin at Weeks 4, 8, 12, 24, 36, and 48;
  Minimum: 0 Maximum: 1 Subjects with a clear(0) or almost clear(1) evaluation were considered PSGA responders.
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 260 | 261
percentage of participants
  Week 4 | 17.1 | 17.2
  Week 8 | 39.3 | 43.7
  Week 12 | 59.1 | 60.7
  Week 24 | 62.4 | 64.7
  Week 36 | 64.6 | 60.8
  Week 48 | 62.4 | 65.5

8. Secondary Outcome: Change in Subject's Global Assessment (SGA) of PsO
Description: Change in Subject's Global Assessment (SGA) of PsO from baseline to Weeks 4, 8, 12, 24, 36, and 48. The SGA of PsO was assessed using VAS (visual analog scale in the unit of millimeters) , ranging from 0 (good) to 100 (severe). The SGA was assessed at randomization (Week 0/Day 0) and Weeks 4, 8, 12, 24, 36, and 48, as well as at the Follow-up Visit, if applicable. The change in SGA is the value at baseline minus sum of values at weeks 4, 8, 12, 24, 36, and 48. Since the change in SGA is measured from baseline, a negative value indicates a decrease in overall SGA and better overall assessment of PsO.
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Population: Part 2 of the study(weeks 13-48) did not include the full analysis population from part 1 of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
units on a scale
  Week 4 | -23.0 (25.11) | -24.0 (22.59)
  Week 8 | -37.1 (25.97) | -35.0 (25.15)
  Week 12 | -45.7 (25.62) | -45.1 (27.81)
  Week 24: number analyzed (Participants) | 213 | 225
  Week 24 | -50.1 (28.50) | -47.2 (28.98)
  Week 36: number analyzed (Participants) | 213 | 225
  Week 36 | -46.9 (29.23) | -47.4 (29.95)
  Week 48: number analyzed (Participants) | 213 | 225
  Week 48 | -50.0 (28.29) | -48.7 (30.12)

9. Secondary Outcome: Change in DLQI (Dermatology Life Quality Index)
Description: Change in DLQI (Dermatology Life Quality Index) from baseline to Weeks 12, 24, and 48
  The DLQI is a 10-question validated questionnaire that was performed at screening, randomization (Week 0/Day 0), and Weeks 12, 24, and 48. It was calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life was impaired.
Time Frame: Weeks 12, 24, and 48
Population: Part 2 (weeks 13-48) of the study did not include the full analysis population from part 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
score on a scale
  Baseline: number analyzed (Participants) | 213 | 225
  Baseline | 17.9 (5.7) | 18.6 (5.86)
  Week 12 | -12.7 (6.2) | -13.4 (7.18)
  Week 24: number analyzed (Participants) | 213 | 225
  Week 24 | -14.3 (6.24) | -14.4 (6.85)
  Week 48: number analyzed (Participants) | 213 | 225
  Week 48 | -13.9 (6.32) | -14.3 (6.81)

10. Secondary Outcome: Change in EuroQol 5-Dimension Health Status Questionnaire (EQ-5D)
Description: Change in EuroQol 5-Dimension Health Status Questionnaire (EQ-5D) from baseline to Weeks 12, 24, and 48
  The EQ-5D was performed at randomization (Week 0/Day 0), and Weeks 12, 24, and 48. The EQ-5D is a generic (non-disease specific), preference-based health-related quality of life measure based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Time Frame: Weeks 12, 24, and 48
Population: Part 2 (weeks 13-48) of the study did not include the full analysis population from part 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
units on a scale
  Week 12 - Mobility | -0.3 (0.81) | -0.3 (0.83)
  Week 12 - Self Care: number analyzed (Participants) | 213 | 225
  Week 12 - Self Care | -0.2 (0.70) | -0.3 (0.73)
  Week 12 - Usual Activities: number analyzed (Participants) | 213 | 225
  Week 12 - Usual Activities | -0.6 (0.94) | -0.4 (0.91)
  Week 12 - Pain/Discomfort: number analyzed (Participants) | 213 | 225
  Week 12 - Pain/Discomfort | -0.9 (1.12) | -0.9 (1.1)
  Week 12 - Anxiety/Depression: number analyzed (Participants) | 213 | 225
  Week 12 - Anxiety/Depression | -0.6 (1.01) | -0.7 (1.01)
  Week 24 - Mobility: number analyzed (Participants) | 213 | 225
  Week 24 - Mobility | -0.3 (0.93) | -0.3 (0.80)
  Week 24 - Self Care: number analyzed (Participants) | 213 | 225
  Week 24 - Self Care | -0.2 (0.70) | -0.3 (0.75)
  Week 24 - Usual Activities | -0.6 (0.96) | -0.5 (0.93)
  Week 24 - Pain/Discomfort: number analyzed (Participants) | 213 | 225
  Week 24 - Pain/Discomfort | -1.0 (1.12) | -0.9 (1.08)
  Week 24 - Anxiety/Depression: number analyzed (Participants) | 213 | 225
  Week 24 - Anxiety/Depression | -0.7 (1.10) | -0.7 (1.06)
  Week 48 - Mobility: number analyzed (Participants) | 213 | 225
  Week 48 - Mobility | -0.4 (0.84) | -0.3 (0.90)
  Week 48 - Self Care: number analyzed (Participants) | 213 | 225
  Week 48 - Self Care | -0.3 (0.70) | -0.3 (0.76)
  Week 48 - Usual Activities: number analyzed (Participants) | 213 | 225
  Week 48 - Usual Activities | -0.7 (0.95) | -0.4 (0.98)
  Week 48 - Pain/Discomfort: number analyzed (Participants) | 213 | 225
  Week 48 - Pain/Discomfort | -1.0 (1.18) | -0.8 (1.13)
  Week 48 - Anxiety/Depression: number analyzed (Participants) | 213 | 225
  Week 48 - Anxiety/Depression | -0.7 (1.08) | -0.6 (1.16)

11. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI - Scales for each question range from 0-3 (0=without any difficulty; 1=with some difficulty; 2=with much difficulty; 3=Unable to do). The "total" for each category is determined by the highest score (greatest difficulty) for that category. The score for the disability index is the mean of the eight category scores. If more than 2 of the categories or 25% are missing, the scale won't be scored. If fewer than 2 or the categories are missing, the sum of the categories was divided by the number of answered categories.
Time Frame: Weeks 12, 24, and 48
Population: Part 2 of the study(weeks-13-48) did not include the full analysis population from part 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
units on a scale
  Week 12 | -0.4 (0.59) | -0.4 (0.39)
  Week 24: number analyzed (Participants) | 213 | 225
  Week 24 | -0.4 (0.75) | -0.5 (0.42)
  Week 48: number analyzed (Participants) | 213 | 225
  Week 48 | -0.6 (0.69) | -0.4 (0.59)

12. Secondary Outcome: Change in Highly Sensitive C-reactive Protein (Hs-CRP; mg/L)
Description: Change in highly sensitive C-reactive protein (hs-CRP; mg/L) from baseline to Weeks 12, 24, and 48 for subjects with PsA (Psoriatic arthritis) only.
  Highly sensitive C-reactive protein For subjects with PsA, change in hs-CRP from baseline to Weeks 12, 24, and 48 was assessed.
Time Frame: Weeks 12, 24, and 48
Population: The population from part 2(weeks 13-48) did not include the full analysis population from part 1.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 228 | 228
mg/L
  Baseline | 11.8 (29.80) | 6.2 (8.39)
  Week 12 | -8.9 (32.10) | -3.3 (6.63)
  Week 24: number analyzed (Participants) | 213 | 225
  Week 24 | -9.1 (31.98) | -1.3 (9.69)
  Week 48: number analyzed (Participants) | 213 | 225
  Week 48 | -11.2 (33.69) | -2.8 (6.01)

13. Secondary Outcome: The Proportion of Subjects With a Durability of Response at Week 48
Description: The proportion of subjects with a durability of response during Part 2. Durability of response was defined as the maintenance of the PASI-50 or greater at Weeks 24, 36, and 48 when compared to baseline (Week 0).
Time Frame: Weeks 24, 36, and 48 when compared to baseline (Week 0).
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 213 | 225
percentage of participants
  Durability of Response - Yes | 77 | 77.8
  Durability of Response - No | 23 | 22.2

ADVERSE EVENTS:
Arm/Group | Enbrel (Etanercept) | CHS-0214
Serious Adverse Events (participants affected / at risk) | 10/260 | 7/261
Other Adverse Events (participants affected / at risk) | 156/260 | 106/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (Etanercept) (N=260) | CHS-0214 (N=261)
Fecaloma (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Esophageal Varices Hemorrhage (Gastrointestinal disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Cardiac Failure (Cardiac disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bartholin's Abscess (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (Etanercept) (N=260) | CHS-0214 (N=261)
Nasopharyngitis (Infections and infestations) | 42 | 40
Upper Respiratory Infection (Infections and infestations) | 27 | 24
Hypertension (Vascular disorders) | 14 | 13
Injection Site Reaction (Injury, poisoning and procedural complications) | 46 | 11
Psoriasis (Skin and subcutaneous tissue disorders) | 14 | 10
Urinary Tract Infection (Infections and infestations) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No